CLINICAL TRIAL: NCT04663425
Title: Is Bariatric Surgery Effective in Super-super Morbid Obese Patients?
Brief Title: Outcome of Bariatric Surgery in Patients With BMI Greater Than 60 .
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of General Surgery Department, Assuta Medical Center
Other Study IDs: AMC-05-20
Record Dates: First submitted 2020-10-16; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-10

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sleeve gastrectomy operation: Outcome of patients that underwent sleeve gastrectomy with BMI greater than 60.
- Gastric bypass operation: Outcome of patients that underwent gastric bypass with BMI greater than 60.
- Gastric Band operation: Outcome of patients that underwent gastric banding with BMI greater than 60.

SUMMARY:
Patients that underwent any type of bariatric surgery with BMI more than 60 will recruited for follow up that includes: actual weight, other surgeries and conversions, co-morbidities status, medications and satisfaction.

DETAILED DESCRIPTION:
Patients that underwent bariatric surgery for BMI =60 or greater were considered for the study. The type of surgery were be analyze related to weight loss. Complication and operation difficulty will be assessed.

Co morbidities and treatment results post surgery will be considered as also, need for revisional surgery/

ELIGIBILITY:
Inclusion Criteria:

BMI above 60 Any bariatric surgery performed including revision

Exclusion Crite ria: Tourist patients Patients under 18 years old

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients accepted to underwent bariatric surgery with BMI equal or above 60
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2008-04-04 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Weight loss after bariatric surgery | from 1 to 12 years
  change in bodyweight following the surgery (kg)
co-morbidities rate following surgery | from 1 to 12 years
  prevalence of diseases linked to obesity (hypertension, diabetes, sleep apnea)